CLINICAL TRIAL: NCT01575002
Title: Neural Correlates of Pain-related Cognitive Processing in Chronic Pain of the Cornea: an ERP and Electrical Stimulation Study.
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) in Chronic Corneal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-p-001902
Record Dates: First submitted 2012-02-08; First posted 2012-04-10 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Corneal Pain; Chronic Pain; Neuropathic Pain
Keywords: transcranial stimulation; direct current stimulation
MeSH Terms: conditions — Chronic Pain; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Subjects will undergo 20 minutes of active tDCS stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Subjects will undergo 20 minutes of sham tDCS stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Subjects will undergo 2 sessions of 20 minutes of tDCS stimulation (either active or sham)in a randomized order - each session will be separated by at least one week to prevent carry-over effects.
  Other Names: 1x1 direct current stimulator; Soterix Medical

SUMMARY:
In this study the investigators aim to examine the effects of Transcranial Direct Current Stimulation (tDCS) on pain levels as well as the changes in cognitive (thought) processing in individuals with chronic pain of the cornea -- and also compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria (for all subjects):

1. Provide informed consent to participate in the study;
2. 18 to 65 years old;

Additional Inclusion Criteria for Subjects with Chronic Corneal Pain:

1. Corneal pain for six months or more;
2. Referral from a corneal specialist (Dr. Perry Rosenthal) with refractoriness to conventional ophthalmologic treatments for corneal pain such as local topical medications and soft bandage contact lenses;
3. Report a Visual Analogue Scale (VAS) for pain of 4 or greater in the previous 3 weeks;

Exclusion Criteria (for all subjects):

1. History of alcohol or substance abuse within the last 6 months as self-reported;
2. Diagnosis of any neurological diseases (such as epilepsy);
3. Episodes of seizures within the last 6 months;
4. Unexplained loss of consciousness
5. Use of carbamazepine or neuropsychotropic drugs
6. Contraindications to tDCS

   * Metal in the head
   * Implanted brain medical devices
7. Pregnant at time of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in pain scales | Measured for approximately 2 weeks
  We will measure changes in the visual analogue scale (VAS) for pain, and also measure pain threshold (using an algometer) before and after each stimulation session. We will compare the measurements from before stimulation to after stimulation, in each scheduled session, as this study is measuring the effects of a single session of tDCS.

SECONDARY OUTCOMES:
Changes in EEG measurements | Measured for approximately 2 weeks
  We will measure changes in event related potentials (ex. P300, mismatch negativity) recorded via electroencephalography (EEG) before and after each stimulation session. We will compare the measurements from before stimulation to after stimulation, in each scheduled session, as this study is measuring the effects of a single session of tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PHD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States